CLINICAL TRIAL: NCT05771649
Title: Differential Effectiveness of Two Recovery Strategies, Based on Mindfulness and Physical Exercise, on Levels of Stress, Academic Performance, and Inmunoglobulin A. A Controlled Trial. A, and Cortisol. A Randomized Controlled Trial
Brief Title: Recovery Strategies Based on Mindfulness and Physical Exercise on Levels of Stress and Inmunoglobulin A
Acronym: ERME-IgA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Educación a Distancia (Other)
Collaborators: Universidad Rey Juan Carlos (Other); Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: PID2019-110490RB-I00 (3)
Record Dates: First submitted 2023-02-22; First posted 2023-03-16 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-02

CONDITIONS: Mental Health Wellness
Keywords: mindfulness; physical exercise; mental health; stress; recovery; Inmunoglobulin A
MeSH Terms: conditions — Motor Activity; Psychological Well-Being | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A non-randomized controlled trial of three groups is proposed, with pretest, posttest and two follow-ups at 1 and 3 months.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding of trial participants and care providers is not possible because of obvious differences between the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness-based intervention (MBI) (Experimental): A 4-week mindfulness-based intervention comprised of focused attention meditations. From 15 to 30 minutes of practice per session, four times/week through audio guides.
  Interventions: Behavioral: Mindfulness-based intervention
- Physical exercise (PE) (Active Comparator): A 4-week physical exercise intervention comprised of running with mental association strategies. From 15 to 30 minutes of practice per session, three times/week through workout audio guides.
  Interventions: Behavioral: Physical exercise
- Treatment as Usual (TAU) (No Intervention): The participants will continue their daily activity and obligations in the academy as usual.

INTERVENTIONS:
Behavioral: Mindfulness-based intervention — A mindfulness instructor will guide focused attention meditations that will last from 15 to 30 minutes. Participants will be instructed at the beginning of the intervention and will have audio files to guide the exercises during their practice.
  Arms: Mindfulness-based intervention (MBI)
Behavioral: Physical exercise — An instructor will guide to running with mental association strategies that will last from 15 to 30 minutes. Participants will be instructed at the beginning of the intervention and will have audio files to guide the exercises during their practice.
  Arms: Physical exercise (PE)

SUMMARY:
The present study aims to compare the differential effects of mindfulness meditation (MBI) and physical exercise (PE) on different stress, academic performance and health variables (self-report means and biological measure of IgA levels). A controlled trial of three groups is proposed, with pretest, posttest and two follow-ups at 1 and 3 months that would be developed among the Guardia Civil (Spanish military police) non-commissioned officers and officers academies.

DETAILED DESCRIPTION:
Recovery from fatigue and daily stress involves mentally disconnecting from the journal. To achieve this disconnection (or psychological detachment), research has shown that engaging in a variety of interesting and motivating activities for individuals after the day allows them to achieve this disconnected state of mind and, consequently, facilitates recovery from work.

Previous research has shown that two of the most effective recovery activities are physical exercise (PE) and mindfulness meditation (MBI), although the results on the differential effects of the two are not conclusive (Karabinski et al, 2021; Steed et al., 2021; Wendsche et al., 2021).

Thus, the present study aims to compare the differential effects of MBI and PE on different stress, academic performance and health variables (self-report means and biological measure of IgA salivary levels). A non-randomized controlled trial (participant chooses to take of three groups proposed) with pretest, posttest and two follow-ups at 1 and 3 months. It would be developed among the Guardia Civil (Spanish military police) non-commissioned officers and officers academies (N ≥ 150). An MBI (focused attention meditations), an aerobic PE program (running with mental association strategies) and an inactive control / waiting list (LE) condition will be contrasted.

The dependent variables considered are: 1) recovery experiences; 2) perceived stress; 3) general health; 4) academic performance; 5) positive and negative affect; 7) daily states of fatigue, stress, psychological distancing, mindfulness, and sleep; 8) IgA levels in saliva. The intervention program is structured for four weeks, during which the two intervention groups will carry out their recovery strategy (MBI or PE), starting and increasing the practice 5 minutes every two weeks. The control group will continue as usual. The investigators believe that this study is a quasi-pioneering initiative because of its theme, and will have an important scientific and technical impact. The importance of the topic addressed in terms of health and academic performance is associated with important contributions in terms of knowledge transfer to the educational field and society in general.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.

Exclusion Criteria:

* Currently practicing any type of meditation regularly.
* To have a physical or mental illness that prevents mindfulness practice.
* To take medication that interferes with salivary inmunoglobulin A (SIgA).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Salivary Immunoglobulin A (SIgA) with four time points data. | Baseline (1 week before interventions), Pre-treatment (the day the interventions start), Post-treatment (4 weeks from the start of the interventions), 1-month follow-up
  Biological measures. Salivary IgA levels as a biomarker of mucosal immunity.
Change in General Health with four time points data. | Pre-treatment (the day the interventions start), Post-treatment (4 weeks from the start of the interventions), 1-month follow-up, 3-month follow-up
  The General Health Questionnaire (GHQ-12) consists of 12 items. It is a unidimensional measure of psychological distress. It is answered on a Likert-type scale from 1 to 4 (1 = Never and 4 = Always). The score was used to generate a total score ranging from 0 to 36. Total scores range from 0 to 36 with a score of 11 or 12 considered typical, scores > 15 suggesting evidence of distress, and scores > 20 are considered severe problems with psychological distress.
Change in stress with four time points data. | Pre-treatment (the day the interventions start), Post-treatment (4 weeks from the start of the interventions), 1-month follow-up, 3-month follow-up
  A single item was used: Stress refers to a person's situation when they feel tense, restless, nervous, or anxious, or are unable to sleep at night because their mind is constantly preoccupied with work-related issues. Please indicate the extent to which you currently feel this type of stress. It has five possible responses on a Likert-type scale from 1 to 5 (being 1 nothing and 5 a lot), with higher scores indicating higher perceived stress
Change in Need for Recovery with four time points data. | Pre-treatment (the day the interventions start), Post-treatment (4 weeks from the start of the interventions), 1-month follow-up, 3-month follow-up
  The Need for Recovery (NFR) Scale consists of 9 items. It facilitates the understanding of the factors that can lead to sustainable working and employability. It is answered on a Likert-type scale from 1 to 5 (1 = Never and 5 = Always).
  The score was used to generate a total score ranging from 1 to 100.Our research team will carry the validation of the Spanish version of NFR. The higher the score, the higher the fatigue symptoms presented by the worker.
Change in Academic Performance with four time points data. | Pre-treatment (grades before the interventions start), 1 and 3-month follow-up (grades after the interventions finish)
  Academic performance will be measured directly through the grades obtained in the academy (by course and by subject).
Change in Positive and Negative Affect with four time points data. | Pre-treatment (the day the interventions start), Post-treatment (4 weeks from the start of the interventions), 1-month follow-up, 3-month follow-up
  The PANAS Scales of Positive and Negative Affect (PANAS) - Spanish version has 20 items. It is the most widely used scale of affectivity. It has two dominant dimensions, positive affect (10 items) and negative affect (10 items) It is answered on a Likert-type scale from 1 to 5 (1 = Very slightly or Not at all and 5 = Extremely). The score was used to generate a total score ranging from 20 to 100. For the total positive score, a higher score indicates more of a positive affect. For the total negative score, a lower score indicates less of a negative affect.

SECONDARY OUTCOMES:
Change in Fatigue (single-item measure from the Single-Item Fatigue Measure) | Time Frame: 4 days per week during the 4-week interventions
  Single-Item on fatigue level:" Indicate what level of fatigue you felt today". The response is recorded on a 5-point Likert scale varying from "not at all" to "very much".
Change in Psychological distancing (item n. 3 from the Recovery Experience Questionnaire). | Time Frame: 4 days per week during the 4-week interventions
  Single-Item on Psychological distancing level: "After work, I have been able to disconnect". The response is recorded on a 5-point Likert scale varying from "not at all" to "very much".
Change in Sleep (item n. 6 from the Pittsburg Sleep Quality Index). | Time Frame: 4 days per week during the 4-week interventions
  Single-Item on Sleep: "How did you sleep last night?". The responses are articulated on a 5-point Likert scale varying from "very bad" to "very good".
Change in Stress (single-item measure from the Single-item Measure of Stress Symptoms). | Time Frame: 4 days per week during the 4-week interventions
  Single-Item on work stress: "Indicate the extent to which you have felt stressed, tense, nervous, or anxious today". The response is recorded on a 5-point Likert scale varying from "not at all" to "very much".
Change in Mindfulness (item n. 3 from the Five Facets Mindfulness Questionnaire). | Time Frame: 4 days per week during the 4-week interventions
  Single-Item on attention: "Today it has been difficult for me to be attentive to what required my attention at all times". The response is recorded on a 5-point Likert scale varying from "not at all" to "very much".

CONTACTS AND LOCATIONS:
Locations (1):
- Raquel Ruiz Iñiguez, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The raw data supporting the conclusions of this article will be made available by the authors, without undue reservation.